CLINICAL TRIAL: NCT04126720
Title: Evaluation of Salivary Total Oxidant Capacity in Oral Lichen Planus Patients Before and After Treatment With Topical Corticosteroid Supplemented With Vitamin E Versus Topical Corticosteroid Alone
Brief Title: Effect of Adjunctive Systemic Vitamin E on Clinical Parameters and Salivary Total Antioxidant Capacity in Symptomatic Oral Lichen Planus Patients: Randomized-controlled Clinical Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Mahmoud Abdel Wahed Abdel dayem, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ED412018
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: No

ARMS (2):
- vitamin E (Active Comparator): topical Corticosteroid (Kenacort A Orabase: triamcinolone acetonide 0.1% 5 gram adhesive paste - Dermapharm) four times daily and Vitamin E capsule (Vitamin E 400: 400 mg vitamin E capsules - Pharopharmaceuticles) daily.
  Interventions: Dietary Supplement: topical corticosteroids and vitamin E suplements
- Placebo (Placebo Comparator): topical Corticosteroid (Kenacort A Orabase: triamcinolone acetonide 0.1% 5 gram adhesive paste - Dermapharm) four times daily and placebo capsule daily
  Interventions: Drug: Topical corticosteroid and placebo capsules

INTERVENTIONS:
Dietary Supplement: topical corticosteroids and vitamin E suplements
  Arms: vitamin E
Drug: Topical corticosteroid and placebo capsules
  Arms: Placebo

SUMMARY:
Treatment of oral lichen planus is challenging. Diverse therapeutic modalities have been suggested, but a permanent cure is not yet available.

In some oral lichen planus patients, topical corticosteroid alone is not sufficiently enough, thus it may require a supplementation to augment its effect.

This trial will assess the effectiveness of vitamin E as a supplement in management of oral lichen planus.

DETAILED DESCRIPTION:
The current study is a randomized-controlled clinical trial that follows CONSORT guideline. The current trial include 30 symptomatic OLP patients in two parallel groups (intervention - topical triamcinolone acetonide adhesive paste and Vitamin E capsule, control - topical triamcinolone acetonide adhesive paste and placebo capsule), with allocation ratio 1:1. Participants were recruited from the pool of the Diagnostic center and the Out-Patient Clinic of Oral Medicine and Periodontology Department, Faculty of Dentistry, Cairo University, Egypt between 2016 and 2017.

This clinical trial followed the principles of the Helsinki Declaration and was approved by the Research ethics committee of Faculty of Dentistry, Cairo University, Egypt (Code: 15733). Each participant was informed about the details of the study and signed a written consent.

Patients were diagnosed clinically and histopathologically (when required). Inclusion criteria included erosive and atrophic OLP patients who agreed to take supplied medications. Exclusion criteria included reticular OLP patients, patients receiving systemic treatment for OLP during the eight weeks prior to the study, patients receiving topical medications for OLP during the four weeks prior to the study, patients suffering from systemic disease; pregnant ladies and lactating ladies.

Interventions:

The intervention was 0.1% triamcinolone acetonide adhesive paste (Kenacort A Orabase - Dermapharm) and 400 mg Vitamin E capsule (Vitamin E 400 - Pharopharmaceuticles) for the experimental group and 0.1% triamcinolone acetonide adhesive paste (Kenacort A Orabase - Dermapharm) and identical placebo capsule for the control group.

Patients were instructed to apply triamcinolone acetonide regularly four times a day after meals and before sleeping for four weeks and to refrain eating and drinking for 30 minutes after the application. In addition, patients were asked to take one capsule (Vitamin E or placebo) once daily at morning.

Outcomes:

Pain intensity was evaluated using numerical rating scale (NRS) at baseline, daily during the first week, then weekly for four weeks. NRS ranges from 0 to 10, with 0 indicating "no pain" and 10 indicating "pain as bad as you can imagine".21 Clinical improvement of the oral lesions was scored using Thongprasom et al. scale at baseline and weekly for four weeks. In Thongprasom et al. scale, lesions are given score as follows: 0, no lesions, normal mucosa; 1, Mild white striae, no erythematous area; 2, White striae with atrophic area < 1 cm2; 3, White striae with atrophic area > 1 cm2; 4, White striae with erosive area < 1 cm2 and 5, White striae with erosive area > 1 cm2.22 Salivary level of TAC was evaluated using ELISA kit. Unstimulated whole saliva samples were used for determination of TAC using ImAnOx (TAS/TAC) Kit provided by Immun Diagnostik, Germany. Participants were asked to refrain eating, drinking or using saliva stimulators for one hour before sample collection. Participants were asked to swallow, then tilt their head forward and expectorate saliva into a centrifuge tubes for 5 minutes without swallowing. The saliva samples were frozen at -70°C, until analysis. The saliva samples were centrifuged at 4500 g for 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically and histopathologically diagnosed as suffering from OLP (erosive and atrophic OLP patients who agreed to take supplied medications).
* Patients free from any visible oral lesions other than OLP.
* Patients who agreed to take supplied medications.
* Patients who agreed for the biopsy

Exclusion Criteria:

* Reticular OLP patients
* Patients suffering from any systemic disease.
* Patients Treated with any systemic treatment such as systemic steroids, other immunosuppressive drugs or non-steroidal anti-inflammatory drugs at least eight weeks.
* Treatment with any oral topical medications for at least four weeks prior to the study.
* Pregnant and lactating mothers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-11-12 (Actual)

PRIMARY OUTCOMES:
Pain measure using numerical rating scale | weekly for 1 month
  All patients will be asked to define their level of pain and discomfort by using a numerical rating scale ranging from 0 to 10 (11-point), with 0 indicating "no pain" and 10 indicating "pain as bad as you can imagine

SECONDARY OUTCOMES:
Clinical improvement of the lesion | weekly for 1 month
  The clinical data will be scored according to the scale used by Thongprasom et al.: 0, no lesions; 1, hyperkeratotic lesions; 2, atrophic area <1 cm2; 3, atrophic area > 1 cm2; 4, erosive area < 1 cm2; 5, erosive area >1 cm2
salivary total anti-oxidant capacity | Preoperative and postoperative
  using the ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No